CLINICAL TRIAL: NCT04445857
Title: Efficacy of Coadministration of Calcitonin and Hyperbaric Bupivacaine in Spinal Anesthesia in Lower Abdominal and Limb Surgeries in Tramadol-abuse Patients: a Randomized Controlled Trial
Brief Title: Efficacy of Coadministration of Calcitonin and Hyperbaric Bupivacaine in Spinal Anesthesia in Tramadol-abuse Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 6379
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): injection of 15 mg (3 ml) hyperbaric bupivacaine 0.5% and 100 IU salmon calcitonin(1ml) intrathecally and injection of 10 ml normal saline (NS) slowly intravenously (IV) over 5 min.
  Interventions: Drug: Calcitonin presented as Miacalcic® ampoules 100 IU/ml (1ml) intrathecally
- Group 2 (Active Comparator): injection of 15 mg (3 ml) hyperbaric bupivacaine 0.5% and 1ml NS intrathecally and injection of 100 IU salmon calcitonin (1ml) diluted in 9 ml NS slowly IV over 5 min.
  Interventions: Drug: Calcitonin presented as Miacalcic® ampoules 100 IU/ml (1ml) intravenously
- Group 3 (control group) (Placebo Comparator): injection of 15 mg (3 ml) hyperbaric bupivacaine 0.5% and 1ml NS intrathecally and injection of 10 ml NS slowly IV over 5 min.
  Interventions: Other: Normal Saline (NS)

INTERVENTIONS:
Drug: Calcitonin presented as Miacalcic® ampoules 100 IU/ml (1ml) intrathecally — coadministration of calcitonin intrathecally and a single-shot hyperbaric bupivacaine
  Arms: Group 1
Drug: Calcitonin presented as Miacalcic® ampoules 100 IU/ml (1ml) intravenously — coadministration of calcitonin intravenously and a single-shot hyperbaric bupivacaine
  Arms: Group 2
Other: Normal Saline (NS) — coadministration of normal saline and a single-shot hyperbaric bupivacaine
  Arms: Group 3 (control group)

SUMMARY:
Increasing duration of local anesthetic action is desired for prolongation of postoperative patient comfort, as well as decreasing perioperative opioid consumption and subsequent side effects. Calcitonin, discovered in 1961, has been established, synthesized, and developed for use in treating disease. In 1983 it was demonstrated that calcitonin is an analgesic, which is also effective in the epidural and subarachnoid spaces.Tramadol abuse has dramatically increased in Egypt since 2008 and has led to many admissions to addiction treatment centers.It was shown that the duration of sensory block of spinal anesthesia with hyperbaric bupivacaine in chronic opium abusers undergoing lower extremity orthopedic surgery was much shorter in chronic opium abusers compared with non-abusers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of tramadol addiction (single drug addiction) and duration of addiction >1 year
* Elective lower abdomen or lower extremities surgeries under spinal anesthesia
* ASA physical status I and II

Exclusion Criteria:

* Patient's refusal,
* duration of surgery more than 120 min,
* obesity with body mass index (BMI) >35 kg/m2,
* generalized infection or localized infection at level of blockade,
* neurological disease,
* psychological disorder
* coagulation disorder,
* history of uncontrolled hypertension,
* history of uncontrolled blood sugar,
* allergy to bupivacaine or calcitonin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The total dose of rescue analgesia (mg) | The first 24 hours after surgery
  The total dose of rescue analgesia (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt